CLINICAL TRIAL: NCT00425399
Title: Shiatsu Adjuvant Therapy for Hospitalized Psychiatric Patients: an Open Pilot Study
Brief Title: Shiatsu Adjuvant Therapy For Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herzog Hospital (Other)
Responsible Party: Dr. Pesach Lichtenberg, Herzog Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lichtenbergCTIL2
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2009-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Shiatsu
MeSH Terms: conditions — Schizophrenia | interventions — Acupressure

INTERVENTIONS:
Procedure: Shiatsu — Shiatsu treatment provided in 40-minute sessions, twice a week for 4 weeks

SUMMARY:
In the current study we will study the effect of adding shiatsu treatment to conventional therapy in work with hospitalized schizophrenic patients.

The hypotheses of this study are several:

1. Shiatsu can improve the patients' symptoms
2. Shiatsu can ameliorate neuromuscular side effects produced by standard anti-psychotic treatment
3. Shiatsu can provide patients with tools to deal with the stresses of their illness

2. Methodology We propose an open pilot study in which a total of 20 patients of both sexes will be enrolled. These patients will be drawn from the inpatient psychiatric wards at Herzog Hospital.

Upon inclusion into the trial, all participants will receive shiatsu treatment, consisting of two individual weekly 40-minute shiatsu treatment sessions for four weeks. Provider and patient will be of the same gender. Standard pharmacotherapy will be provided as needed during the treatment period. Medication and dosage will not be changed. If necessary, benzodiazepines will be administered as required.

Outcome measures:

The following assessments will be included:

1. Medication: Use of SOS benzodiazepines
2. Clinical rating scales: PANSS, CGI, NOSIE, Hamilton Scales for depression and anxiety

1. Side effect scales: Simpson Angus Scale, AIMS scale, UKU scale 2. Neurophysiological testing: Prepulse inhibition (PPI). 3. Neurocognitive testing: This will be performed using the NIMH's Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery for Clinical Trials.

DETAILED DESCRIPTION:
SHIATSU ADJUVANT THERAPY FOR SCHIZOPHRENIA Protocol for an Open Pilot Study

1. Background Schizophrenia is a severe, chronic mental illness that affects approximately 1% of the population worldwide. While the pharmacological treatments available have advanced considerably in the last fifty years, there are limits to what they offer some patients, especially in terms of improving dysphoria, sleep, mood, avolition, social functioning, and anhedonia, which contribute greatly to the everyday misery of these patients.

Furthermore, some of the antipsychotic drugs induce side effects of parkinsonism, akathisias, orofacial dyskinesias, dystonias, and their associated muscle pain, and stiffness. The treatments used for those side effects are anticholinergic drugs (e.g. trihexyphenidyl), benzodiazepines, and beta blockers. The number and variety of such drugs suggests what clinicians know to be unfortunately true: there are no magic bullets for these symptoms. These drugs are also not innocent, causing side effects of their own, contributing to polypharmacy, and carrying a financial cost.

Schizophrenia, then, remains a debilitating illness whose treatment results are often partial and may produce unpleasant side-effects. New approaches to supplement standard modalities ought to be considered.

Shiatsu, or acupressure, is a holistic form of medicine originating in Japan but now widely practiced throughout the world. Shiatsu involves applying pressure to "meridians" of the body, much like acupuncture but without the needles. The shiatsu therapist views the whole body as interconnected - stiffness in one part may reflect a problem in another, or emotional disharmony. In accordance with the WHO definition of health as "a state of complete physical, mental and social well-being and not merely the absence of disease or infirmity," shiatsu massage aims to improve the overall well-being of its recipients by manipulating the body.

Shiatsu theory is based on traditional Chinese medicine, which posits meridians of life force (chi) running through the body, and aims to optimize health through manipulating the body into maximal alignment. Disease, according to this approach, is as an accumulation of damage and stress that causes the body to tense up in various areas, leading to health disturbances. The treatment aims to loosen tense muscles and tendons and restore balance to the body.

Shiatsu also involves a diagnostic process that is designed to locate sources of problems. The main four areas of this process are the patient's appearance, his/her voice, the specific complaints and medical history of the patient, and touch diagnosis. The touch is meant to reveal areas of excess or lack of energy in the body or internal organs and autonomic nervous system. Treatment is individualized according to the findings of this examination.

Goals of treatment, in addition to releasing muscle and tendon tension and protecting these structures, are to help the patient acquire an awareness of his or her body and psyche in order to avoid recurrence of the problems, to identify life stressors (mental and physical), and to strengthen the patient's overall energy flow and resilience to disease.

The two fields of shiatsu are do-in and anma. Do-in are the exercises that involve stretching parts of the body combined with breathing exercises in order to loosen tense joints and improve general circulation. Anma shiatsu is the more familiar massage-type treatment. However, it is not performed for comfort or pleasure, as in Western massage, but rather as a type of medical treatment. It is performed with a fully dressed patient, with direct pressure applied with the practitioner's fingers. Both diagnosis and treatment are performed this way, with the findings of the exam directing further actions.

How might the effects of shiatsu be explained in terms of Western medicine? In order to answer this, we will consider research done not only for shiatsu but for acupuncture as well, which has been more extensively examined. This is justified for two reasons: first of all, shiatsu and acupuncture share the same understanding of human functioning and disease, including the core concepts of chi and meridians, and accordingly they recognize the same points along the body for applying pressure (shiatsu) or needles (acupuncture). Secondly, in studies which have been conducted to test the effectiveness of alternative remedies, acupressure and acupuncture have often been combined (e.g. Vachiramon & Wang, 2005; Melchart et al, 2006).

2. Biological basis for shiatsu Medical research has attempted to understand how Chinese medicine works its effects. Several theories have been developed which may be of relevance to schizophrenia.

1. Endorphins: The most established effect of acupuncture is the release of endorphins, which are endogenous opioid neuropeptides (Hökfelt, 1991; Sjölund et al, 1977). Endorphin release appears to be closely related to the analgesic effects of acupuncture. Endorphins also promote a general feel of well being and reduction of tension which can have salutary effects in treating mental illness.
2. Cytokines: Cytokines mediate the inflammatory response. They also promote endorphin release by the pituitary (Van der Meer et al, 1996). Drzyzga et al (2006) have reviewed the possible connection between cytokines on the one hand, and neuropathological changes, schizophrenia, and anti-psychotic medication mechanisms of action on the other. A growing body of evidence suggests that cytokinins mediate neuropathological changes in schizophrenia and the antipsychotic effects of medication. Acupuncture has been shown to affect the cytokine system in animal (Liu et al, 2004) and human (Petti et al, 2002) studies. The cytokine system is theoretically a pathway through which acupuncture could produce therapeutic effects upon schizophrenia.
3. Glutamatergic mechanisms gained prominence as an important factor in the pathogenesis and treatment of schizophrenia. In experiments with animals, N-methyl-D-aspartic acid (NMDA) receptor antagonists have synergistically enhanced the anti-nociceptive effects of electro-acupuncture (Zhang et al, 2002). Assessing the relationship between glutamatergic activity and acupuncture effects could provide important information about therapeutic mechanisms of action.
4. Neuropeptide Y (NPY): NPY's role in the CNS is not well understood. However, appreciation for the possible role of NPY in the pathogenesis of severe mental disorder has increased in recent years. NPY mRNA levels were significantly reduced in the frontal cortex of patients with both schizophrenia and bipolar disorder (Kuromitsu et al, 2001). NPY has also been shown to play a role in mediating the effects of antipsychotic medication, in both animal (Huang et al, 2006) and human studies (Obuchowicz et al, 2004). Interestingly, the effects of NPY may be mediated by glutamatergic mechanisms (Rosse & Deutsch, 2004). This is relevant to our study because NPY levels in saliva have been found to increase following acupuncture treatment (Dawidson et al, 1998). This, then, is another possible mechanism through which acupuncture can be clinically relevant to the treatment of schizophrenia.

Studies have already been carried out to assess the effectiveness of Chinese medicine in the treatment of schizophrenia. In a recent review of five studies in the Cochrane Database (Rathbone & Xia, 2005), acupuncture as adjuvant therapy provided with anti-psychotic medication showed some evidence of improved outcomes on clinical rating scales and side effect profiles, though overall the evidence was deemed insufficient to reach a definite conclusion, and "more comprehensive and better designed studies" were recommended.

A second review (Moffet, 2006) of clinical trials of acupuncture for various medical disorders made the important observation that too often, no meaningful physiological rationale is provided for the proposed effectiveness of the treatment. Proposing a rationale enables the investigator to suggest a testable causal hypothesis which can contribute to our knowledge of the technique's mechanism of action.

In the current study we will focus on assessments of the glutamatergic system by neurophysiological (prepulse inhibition) testing using prepulse inhibition (PPI). In this paradigm, the subject is presented with an auditory stimulus, or "pre-pulse", which would not ordinarily cause the subject to blink. Following this initial prepulse by a tenth of a second comes a second, louder stimulus, the pulse, which would cause blinking were it not preceded by the prepulse. Pre-pulse inhibition, a measure of sensory gating or filtering, is determined by the reduction in blink response to a pulse following a pre-pulse as compared to the blink response without the preparatory pre-pulse. Prepulse inhibition of the startle response, which has been reliably demonstrated in both humans and animals (rev. in Braff et al., 2001; Swerdlow et al., 2001), is a preattentive, automatic process.

Schizophrenia patients have been repeatedly shown reduced inhibition of the startle reflex in PPI (rev. in Geyer et al., 2001). This loss of normal PPI is thought to be a measure of the deficient sensorimotor gating (Braff and Geyer, 1990) that underlies sensory flooding and cognitive fragmentation in these patients (McGhie and Chapman, 1961). Furthermore, some studies report that PPI deficits may correlate with symptoms severity or cognitive and functional impairment in schizophrenia and may partially or completely resolve with antipsychotic drugs treatment (rev. in Braff et al., 2001).

One of the proposed models of PPI hypothesizes the involvement of glutamatergic, mainly N-methyl-D-aspartate receptor (NMDAR)-mediated neurotransmission. Glutamate is a key inhibitory neurotransmitter. Glutamatergic neurotransmission may correlate with the efficiency of sensory gating (Swerdlow and Geyer, 1999). Glutamatergic synapses have been implicated in the regulation of PPI in rodents (Swerdlow et al., 2001).

In light of the possible connection between PPI and the glutamatergic system, we decided to administer PPI to the subjects before and after the shiatsu treatment in order to assess whether any ameliorating effect of shiatsu, which as noted can involve glutamatergic mechanisms, may correlate with changes in the PPI.

We will also assess neurocognitive function using a battery of tests developed specifically for use in assessing patients with schizophrenia.

3. Study goals: Based upon the rationales we suggested for utilizing shiatsu in the treatment of schizophrenia, and based upon the studies which have already been performed, we are proposing a pilot study to examine the efficacy of shiatsu as adjuvant therapy for antipsychotics in the treatment of patients with schizophrenia.

The goals of this study are several:

1. To improve the patients' symptoms 2. To ameliorate neuromuscular side effects produced by standard anti-psychotic treatment 3. To provide patients with tools to deal with the stresses of their illness 4. To provide a basis for further investigation of the effects of shiatsu 4. Methodology We propose an open pilot study in which a total of 20 patients will be enrolled. These patients will be drawn from the inpatient psychiatric wards at Herzog Hospital. They will be recruited by the treating physicians at these facilities. All patients would be fully informed of the experimental treatments, goals, and possible outcomes. Either the participant, or where relevant the court-appointed guardian, will be required to provide informed consent. Participants will of course be free to discontinue their participation for any reason at any time.

4.1 Inclusion Criteria:

1. DSM-IV-R diagnosis of schizophrenia or schizoaffective disorder
2. Ages 18 and over
3. Clinical status stable, as reflected by at least one month of drug treatment without change of anti-psychotic drug or dosage.
4. Ability to cooperate with 40-minute sessions 4.2 Exclusion Criteria:

<!-- -->

1. Active fracture or other orthopedic problem
2. Skin condition that renders treatment unsafe or painful
3. Active infection in skin or soft tissues, such as cellulitis
4. Any acute illness or other medical condition (e.g. solid tissue malignancy) for which shiatsu may be contraindicated.

4.3 Study design Upon inclusion into the trial, all participants will receive shiatsu treatment, consisting of two individual weekly 40-minute shiatsu treatment sessions for four weeks. The shiatsu providers are all trained and certified by Tsabar College, an alternative medicine training institute, and all have at least two years of post-training experience in shiatsu. Each patient will receive all treatments from the same provider for the duration of his or her treatment. Provider and patient will be of the same gender. The patient is clothed with a shirt and full-length trousers or skirt during shiatsu. Treatment will not include contact with sensitive regions of the body, such as the chest (in work with females), pelvic, or inner thigh regions, or any other region of the body with which the patient is not comfortable.

Standard pharmacotherapy will be provided as needed during the treatment period. Medication and dosage will not be changed. If necessary, benzodiazepines will be administered as required.

4.4 Rescue strategies and withdrawal from research In case of exacerbation, defined as an increase of 2 points on the BPRS (or 4 to 6 on the individual items listed above), or of one point on the CGI, the patient may receive clothiapine at a dose of up to 80 mg/day for not more than 3 days within a 14-day period.

In case of relapse, defined as an increase of 3 points on the BPRS (or from 5 to 7 on somatic concern, conceptual disorganization, hostility, suspiciousness, hallucinatory behavior or unusual thought content), or of 2 points on the CGI, the patient will be withdrawn from the study and appropriate treatment instituted. Furthermore, if the patient deteriorates clinically in a way that may be related to treatment (e.g. paranoid fantasies directed towards the shiatsu therapist), the research protocol for that individual will be discontinued.

Significant emergent medical problems will also lead to the withdrawal of the patient from the research.

4.5 Outcome measures

The following assessments will be included:

1. Medication

   a. Use of SOS benzodiazepines: quantity and frequency
2. Clinical rating scales

   1. PANSS
   2. CGI
   3. NOSIE
   4. Hamilton Scales for depression and anxiety

2. Side effect scales:

1. Simpson Angus Scale
2. AIMS scale
3. UKU scale 3. Neurophysiological testing: Prepulse inhibition (PPI). This is performed as follows: The eyeblink component of the acoustic startle reflex is measured using electromyography of the obicularis oculi muscle. Two electrodes (6 mm) Ag/AgCl electrodes filled with electrode gel (parker laboratories inc.) will be positioned below and to the right of the patient's right eye, over the obicularis oculi muscle. Electrodes will be placed to minimize potential electro-oculogram artifact. Specifically, 1 electrode will be placed approximately 1 cm lateral to and 0.5 cm below the lateral canthus, and the second electrode will be placed approximately 1.5 cm below and slightly medial to the first electrode, conforming to the location of the obicularis oculi fibers. A ground electrode will be placed behind the right ear over the mastoid. All resistances will be less than 10 kOhm. Electrodes will be fixed to the skin as close as possible to each other using adhesive collars. All acoustic stimuli will be delivered binaurally through headphones (Maico, TDH-39-P). Subjects will be seated comfortably in a softly lit after they will be informed of the procedure. The prepulse and startle stimuli are bursts of white noise with a fixed interstimulus intervals of 30, 60 and 120 ms for measuring PPI or 15 ms and 4500 ms for measuring PPF. The startle session will begin with a 5-minute acclimation period of 70-dB white noise, which will continue throughout the session, followed by six trial blocks. Block 1 consisted of six pulse-alone trials. Blocks 2 and 3 each consisted of 32 trials, containing 8 pulse-alone and 24 prepulse-pulse trials presented in pseudorandom order. Block 4 consisted of six pulse-alone trials. Block 5 consisted of six pulse-alone trials and 12 prepulse-pulse trials and block 6 consisted six pulse alone trials. The first, forth and sixth blocks will measure habituation as well as startle response, the second and the third blocks will measure startle response and PPI and the fifth block will measure PPF. The pulse alone stimulus is a 40 ms presentation of 115dB white noise, the prepulse stimulus is a 20 ms (except the 15 ms interval stimulus which lasts 5 ms) presentation of 86 dB noise, both over 70 dB of continuous background noise. Acoustic stimuli consist of pulse alone, prepulse and pulse, or no stimulus trials and are presented in a fixed pseudorandom order. Electromyographic activity recorded by the electrodes will be directed through a customized electromyographic amplifier to a computerized startle response monitoring system for digitization and analysis (SR-LAB; San Diego Instruments Inc, San Diego, Calif). The system will record 1000 one-ms readings starting at the onset of the startle stimulus. Acoustic startle and prepulse stimuli will be presented binaurally through headphones.

   4. Neurocognitive testing: This will be performed using the NIMH's Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery for Clinical Trials. This recently-developed battery is recommended for use in clinical trials of putative cognition-enhancing agents in schizophrenia. The MATRICS battery, including Hebrew translations of relevant tests, is presently used in the Stanley Foundation-sponsored Israel Multicenter D-Serine Trial (IMSER) (Dr. Heresco-Levy - Co-Principal Investigator) and will be implemented by a trained psychologist presently participating in this project.

   5. Hypothesis: Shiatsu adjuvant therapy will improve psychiatric and motor symptoms in patients after four weeks of therapy.

   6.1 Potential Benefits: Shiatsu treatment is a pleasant experience involving applying pressure manually to various points of the body. Furthermore, the research will itself lead to more time spent by staff with patients, which is to the patient's benefit. Beyond that we anticipate that shiatsu will be of benefit, alongside the standard pharmacological treatment which will be continued, in enhancing the patient's wellbeing and reducing medication side effects.

   6.2 Potential Adverse Effects: Shiatsu is not known to carry any significant risks to patients. It may rarely cause soreness, muscle cramps, or local pain. Patients will be informed of this possibility and instructed to notify the shiatsu therapist if discomfort occurs during treatment. Psychological distress may be aroused by the human contact and touching that occurs during treatment. Patients will be advised about this possibility as well. Patients wishing for any reason to discontinue the research will of course be withdrawn from the study.

   6.3 Significance of study: The treatment of schizophrenia could benefit from new modalities to complement existing approaches. To date, no study has systemically evaluated the use of shiatsu in treating schizophrenia, and only one study has evaluated shiatsu in this population for drug induced myospasm. Due to the chronic nature of this disease and the severe impairment of quality of life, any and all means should be sought in combating the suffering inherent in this disease. Shiatsu may be a cost-effective, pleasant, and well-tolerated treatment for some schizophrenia symptoms. This study may pave the way for similar studies in other psychiatric patients.

   7. References Braff DL, Geyer MA. (1990). Sensorimotor gating and schizophrenia: human and animal model studies. Archives of General Psychiatry 47, 181-188.

   Braff DL, Geyer MA, Swerdlow NR. (2001). Human studies of prepulse inhibition of startle: normal subjects, patient groups, and pharmacological studies. Psychopharmacology 156, 234-258.

   Dawidson I, Angmar-Månsson B, Blom M, Theodorsson E, Lundeberg T. The influence of sensory stimulation acupuncture on the release of neuropeptides in the saliva of healthy subjects. Life Sciences 1998, 63: 659-674 Drzyzga L, Obuchowicz E, Marcinowska A, Herman ZS. Cytokines in schizophrenia and the effects of antipsychotic drugs. Brain Behav Immun. 2006 Geyer MA, Krebs-Thomson K, Braff DL, Swerdlow NR. (2001). Pharmacological studies of prepulse inhibition models of sensorimotor gating deficits in schizophrenia: a decade in review. Psychopharmacology 156, 117-154.

   Hökfelt T. Neuropeptides in perspective: the last ten years. Neuron 1991; 7: 867±879.

   Huang XF, Deng C, Zavitsanou K.Neuropeptide Y mRNA expression levels following chronic olanzapine, clozapine and haloperidol administration in rats. Neuropeptides. 2006 Jun;40(3):213-9.

   Liu XY, Zhou HF, Pan YL, Liang XB, Niu DB, Xue B, Li FQ, He QH, Wang XH, Wang XM. Electro-acupuncture stimulation protects dopaminergic neurons from inflammation-mediated damage in medial forebrain bundle-transected rats. Exp Neurol. 2004 ;189(1):189-96.

   McGhie A, Chapman J. (1961). Disorders of attention and perception in early schizophrenia. British Journal of Medical Psychology 34, 102-116.

   Melchart D, Ihbe-Heffinger A, Leps B, von Schilling C, Linde K. Acupuncture and acupressure for the prevention of chemotherapy-induced nausea--a randomised cross-over pilot study. Support Care Cancer. 2006 Aug;14(8):878-82.

   Moffet HH. How might acupuncture work? A systematic review of physiologic rationales from clinical trials. BMC Complementary and Alternative Medicine 2006; 6: 25-32.

   Obuchowicz E, Krysiak R, Herman ZS. Does neuropeptide Y (NPY) mediate the effects of psychotropic drugs? Neurosci Biobehav Rev. 2004 Oct;28(6):595-610.

   Petti FB, Liguori A, Ippoliti F. J Tradit Chin Med. Study on cytokines IL-2, IL-6, IL-10 in patients of chronic allergic rhinitis treated with acupuncture. 2002;22(2):104-11.

   Rathbone J, Xia J. Acupuncture for schizophrenia. Cochrane Database Syst Rev. 2005 ;(4):CD005475.

   Rosse RB, Deutsch SI. The "Yoking" of glutamatergic brain mechanisms involved in controlling brain neuronal excitability and psychosis to brain mechanisms involved in appetite regulation: a new hypothesis on the origin of psychosis. Med Hypotheses. 2004;62(3):406-12.

   Sjölund B., Terenius L., Erickson M. Increased cerebrospinal fluid levels of endorphins after electro-acupuncture. Acta Physiol Scand 1977; 100: 382±384.

   Swerdlow NR, Geyer MA. (1999). Neurophysiology and neuropharmacology of short lead interval startle modification. In: Dawson ME, Schell AM (Eds.), Startle Modification: Implications for Neuroscience, Cognitive Science, and Clinical Science (pp. 114-133), New York: Cambridge University Press.

   Swerdlow NR, Geyer MA, Braff DL. (2001). Neural circuitry of prepulse inhibition of startle in the rat: current knowledge and future challenges. Psychopharmacology 156, 1940-215.

   Vachiramon A, Wang WC. Acupuncture and acupressure techniques for reducing orthodontic post-adjustment pain. J Contemp Dent Pract. 2005; 6(1):163-7.

   Van der Meer M. J., Hermans A. R., Pesman G. J., Sweep C. G. Effect of cytokines on pituitary beta endorphin and adrenal corticosterone release in vitro. Cytokine 1996; 8: 238±247.

   Zhang YQ, Ji GC, Wu GC, Zhao ZQ. Excitatory amino acid receptor antagonists and electroacupuncture synergetically inhibit carrageenan-induced behavioral hyperalgesia and spinal fos expression in rats. Pain. 2002;99(3):525-35.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-R diagnosis of schizophrenia or schizoaffective disorder
2. Ages 18 and over
3. Clinical status stable, as reflected by at least one month of drug treatment without change of anti-psychotic drug or dosage.
4. Ability to cooperate with 40-minute sessions

Exclusion Criteria:

1. Active fracture or other orthopedic problem
2. Skin condition that renders treatment unsafe or painful
3. Active infection in skin or soft tissues, such as cellulitis
4. Any acute illness or other medical condition (e.g. solid tissue malignancy) for which shiatsu may be contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-01; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pesach Lichtenberg, M.D., Principal Investigator — Herzog Hospital
Locations (1):
- Herzog Hospital, Department of Psychiatry, Jerusalem, Israel